CLINICAL TRIAL: NCT05530044
Title: Developing and Evaluating Messaging Strategies to Increase Peer Education About COVID-19 Vaccination and Climate Change Among Adults in the United States
Brief Title: Messaging Strategies to Increase Peer Education on COVID-19 Vaccination and Climate Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00018956
Record Dates: First submitted 2022-08-31; First posted 2022-09-07 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Vaccine Hesitancy; Climate Change
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: online
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaccine (Experimental): Promotes COVID-19 vaccine uptake
  Interventions: Behavioral: Social diffusion intervention
- climate change (Active Comparator): Promotes climate change activism
  Interventions: Behavioral: Social diffusion intervention

INTERVENTIONS:
Behavioral: Social diffusion intervention — training in communication skills

SUMMARY:
The primary objective of this protocol is to develop and evaluate peer communication interventions to encourage peer education around COVID-19 vaccination and climate change.

DETAILED DESCRIPTION:
Investigators will use a RCT peer education intervention to address climate change-related behaviors as a control condition for the vaccination intervention. Both issues represent serious public health priorities and are sufficiently unrelated in order to act as control conditions for each other.

As a control topic, investigators will address climate change communication. This parallel topic was selected because it is (1) reasonably unrelated to the COVID-19 condition, (2) has clear individual-level behaviors that can be targeted for intervention, (3) has diversity in public attitudes like COVID-19 vaccines,18 (4) has parallels in COVID-19 in terms of polarization and discrediting of scientific research, (5) represents a significant threat to population health, and (6) has significant racial and ethnic disparities paralleling those of COVID-19.

Investigators will recruit a second sample of up to 800 eligible participants who will be asked to complete an intervention session, where they will receive training on how to talk to members of their social network about either COVID-19 vaccination or climate change. The two intervention conditions will differ based on topic (vaccination/climate change) but the intervention components will be comparable. During the intervention, participants will watch a series of videos that teach key communication skills for having conversation about the assigned topic. Additional videos will provide training in how to use social media as a communication platform to share information in case participants are unfamiliar. Participants will then complete practice activities where they will construct hypothetical conversations and react to/critique example conversations to practice implementing the communication skills. Upon completing the intervention, participants will be asked to try to talk to others in their social network about the topic area they were assigned to.

Two to four weeks after the intervention, participants who completed the intervention will be asked to complete a follow-up survey to assess whether participants had conversations with others in their social networks, if they used social media/text/e-mail to share accurate information, and to understand the outcome of the conversations (i.e. did they result in behavior change).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* English-reading
* Reside in the United States
* Over 18 years of age
* Have passed Prolific's data quality checks on their previously submitted work
* Have heard of COVID-19 and the COVID-19 vaccine

Exclusion Criteria:

* Do not provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Frequency of conversations about vaccines | 1 month
  A brief measure of frequency of conversations about vaccines in the prior month
Frequency of conversations about climate change | 1 month
  A brief measure of frequency of conversations about climate in the prior month
Actions to promote vaccine uptake in social network | 1 month
  Number of social network members that participate encouraged to become vaccinated
Actions to promote climate change activism in social network | 1 month
  Number of social network members that participate encouraged to engage in climate change actions

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Latkin, Ph.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
unidentified data
Supporting Information: Study Protocol, ICF
Time Frame: Two years from the end of the study.
Access Criteria: contact the PI.